CLINICAL TRIAL: NCT07405671
Title: Randomized Evaluation of fleCAinide Safety Versus STandard of Care in Patients With Coronary Artery Disease and Atrial Fibrillation
Brief Title: Flecainide Safety in Patients With Coronary Artery Disease and Atrial Fibrillation
Acronym: ReCAST AF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S69367; 2025-525121-13 (EudraCT Number)
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Coronary Artery Disease
Keywords: atrial fibrillation; rhythm control; stable coronary artery disease; flecainide; sotalol; amiodarone
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — Flecainide; Sotalol; Amiodarone

STUDY DESIGN:
Intervention Model Description: Multicenter, pragmatic, 2-arm, parallel group, open-label, individually randomised controlled non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flecainide (Experimental): Flecainide, a class Ic anti-arrhythmic drug.
  Interventions: Drug: flecainide
- Sotalol or Amiodarone (Active Comparator): Class III anti-arrhythmic drug: sotalol or amiodarone as per physician preference.
  Interventions: Drug: Sotalol or Amiodarone

INTERVENTIONS:
Drug: flecainide — Flecainide, a class Ic anti-arrhythmic drug Recommended starting dose of 100 to 150 mg per day per os, either spread in 2 equal doses BID or in 1 dose OD with controlled release formulation.
  Flecainide will always be combined with an AV nodal blocker (beta-blocker or diltiazem/verapamil).
  Arms: Flecainide
Drug: Sotalol or Amiodarone — Class III anti-arrhythmic drug: Sotalol or amiodarone as per physician preference.
  Recommended starting doses:
  * Sotalol: 80 mg BID per os, with a dose adjustment to once daily if the eGFR is between 40 and 60 mL/min.
  * Amiodarone: loading dose of 600 mg daily per os in divided doses for 1 week, followed by 400 mg daily per os in divided doses for 1 week, and subsequently 200 mg per os once daily.
  Arms: Sotalol or Amiodarone

SUMMARY:
The goal of this clinical trial is to learn whether the antiarrhythmic drug flecainide can be used as safely as standard rhythm-control drugs in people with atrial fibrillation (AF) and stable coronary artery disease (CAD). The study includes adults aged 18 years and older who have AF and known but stable coronary artery disease.

The main questions this study aims to answer are:

* Is treatment with flecainide as safe as standard rhythm-control drugs (sotalol or amiodarone) in this patient group?
* Does flecainide lead to similar or fewer serious side effects, hospitalisations, or deaths compared with standard treatment?

Researchers will compare patients treated with flecainide to patients treated with standard rhythm-control therapy (sotalol or amiodarone) to see whether flecainide is not worse in terms of safety outcomes.

Participants will:

* Be randomly assigned to receive either flecainide or standard rhythm-control medication
* Take the assigned medication as part of routine clinical care
* Attend regular follow-up visits at the hospital and have additional follow-up by telephone
* Undergo routine heart tests such as electrocardiograms and echocardiography
* Complete questionnaires about symptoms, quality of life, and daily functioning

This study follows patients for at least one year and collects information on safety, heart rhythm outcomes, quality of life, and healthcare use.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form
3. Non-permanent atrial fibrillation or ectopic atrial tachycardia with rhythm control strategy, documented on any modality in the 1 year preceding the consent date
4. Stable coronary artery disease without argument, defined as:

   1. Prior percutaneous coronary intervention; OR
   2. Prior revascularised ACS or coronary artery bypass surgery > 3 months at enrolment; OR
   3. Invasive coronary angiography demonstrating coronary atherosclerosis, defined as ≥50% diameter stenosis in at least one major epicardial coronary artery; OR
   4. Coronary CT scan showing coronary stenosis CAD-RADS stage ≥ 3 on, including CAD-RADS stages 4 and 5 in the absence of ischemia on exercise testing, myocardial perfusion imaging (MIBI), stress cardiac MRI, or fractional flow reserve.
5. LVEF ≥ 45% documented on any imaging modality*

Exclusion Criteria:

1. LVEF < 45%
2. NYHA class III or IV congestive heart failure
3. Active treatment with amiodarone
4. History of intolerance of flecainide or both sotalol and amiodarone
5. Unstable angina or inducible ischemia on exercise stress testing, myocardial perfusion imaging, stress cardiac MRI, or fractional flow reserve performed for clinical indications
6. Baseline QRS duration ≥ 120 ms, unless a functioning pacemaker is present
7. Baseline corrected QT interval (Fridericia) ≥ 500 ms
8. Pre-existing advanced AV block (second-, or third-degree)
9. Pre-existing sick sinus syndrome or sinus bradycardia <50 bpm
10. Known channelopathy
11. Contra-indication to AV-slowing agents, including beta-blockers, diltiazem or verapamil
12. Atrial fibrillation due to reversible cause
13. Active intracardiac thrombus
14. Acute coronary syndrome during the 3-month period preceding the consent date
15. Cardiac surgery, including coronary artery bypass surgery, during the 3-month period preceding the consent date or planned at a future date at the time of consent
16. Moderate or severe congenital heart disease as per 2020 ESC guidelines
17. Hypertrophic cardiomyopathy (septal or posterior wall thickness >1.5 cm)
18. Significant chronic kidney disease (eGFR <40 mL/min)
19. Life expectancy less than 1 year
20. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate, highly effective contraceptive
21. Inability to provide written informed consent, including decision-making incapacity due to cognitive impairment or other medical or psychiatric conditions that preclude adequate understanding of the study and its procedures.
22. Participation in an interventional Trial with an investigational medicinal product (IMP) or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 988 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Composite safety outcome | 1 year
  The primary outcome measure is a composite safety outcome including all-cause mortality, severe adverse events leading to drug discontinuation, and unscheduled hospitalisation for heart failure or acute coronary syndrome. Each of these individual components is assessed as secondary outcome.

SECONDARY OUTCOMES:
All-cause mortality | 1 year
  Death from any cause
Severe adverse events leading to drug discontinuation | 1 year
  Any severe AE leading to intervention discontinuation, including bradyarrhythmias, ventricular arrhythmias, atrial flutter with 1:1 conduction, QT/QRS prolongation, serious extra-cardiac adverse events
Unscheduled hospitalisation for heart failure or acute coronary syndrome | 1 year
  Unscheduled hospitalisation for heart failure or acute coronary syndrome
AF recurrence | 1 year
  Freedom from fast atrial arrhythmia post-treatment (clinical recurrence of AF)
Major adverse cardiovascular events | 1 year
  Composite of cardiovascular death, myocardial infarction, stroke
Catheter ablation | 1 year
  Incidence of catheter ablation for AF during follow-up
Cardiovascular hospitalisation duration | 1 year
  Total number of days of cardiovascular hospitalisation
Treatment-related adverse events | 1 year
  All serious adverse events and adverse events:
  * Frequency and severity of all treatment-emergent adverse events
  * Proportion of participants experiencing at least one AE/SAE.
  * Specific drug-related adverse events (e.g., QT prolongation, proarrhythmia, bradycardia, hypotension, fatigue, gastrointestinal disturbances).
Cardiac function - LVEF | 3 months
  Changes in cardiac function assessed by left ventricular ejection fraction expressed in percentages (%) from baseline measured by echocardiography
NT-proBNP | 3 months
  Change in N-terminal-pro-brain Natriuretic Peptide (NT-proBNP) at 3 months from baseline
QTc | 1 year
  Change in QTc interval (ms) and QRS duration (ms) from baseline
Healthcare resource utilization | 1 year
  Total within-trial healthcare resource utilization expressed in Euro (€)
Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire | 1 year
  Change in patient reported outcomes assessed by the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire. The AFEQT questionnaire is a 20-item, disease-specific, patient-reported outcome measure ranging from 0 to 100 with a higher value corresponding to a better quality of life.
EuroQoL-5 dimension health utility index (EQ-5D-5L) | 1 year
  Change in patient-reported outcome as assessed by the EuroQoL-5 dimension health utility index (EQ-5D-5L) questionnaire. The EQ-5D-5L measures health-related quality of life across five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) on five severity levels (1=no problem to 5=extreme problem). Results are interpreted via a 5-digit health state profile (e.g., 11211), a calculated utility index (ranging from <0 to 1, where 1=full health), and a 0-100 Visual Analog Scale (VAS). A higher score corresponds to a better quality of life.
Short Form-12 (SF-12) health survey | 1 year
  Change in patient-reported outcome as assessed by the Short Form-12 (SF-12) health survey. The Short Form-12 (SF-12) health survey is interpreted by calculating two main, norm-based scores-the Physical Component Summary (PCS) and Mental Component Summary (MCS)-where a score of 50 represents the average for the general population. Scores above 50 indicate better-than-average health-related quality of life, while scores below 50 indicate below-average health.
EHRA symptom score | 1 year
  Change in patient-reported outcome as assessed by the European Heart Rhythm Association (EHRA) symptom score. The EHRA symptom score is a standardized, four-level classification system used to quantify the severity of symptoms in patients with atrial fibrillation based on how they impact daily activities.
  EHRA Symptom Score Classification (I-IV):
  EHRA I (Asymptomatic): No symptoms are experienced. EHRA II (Mild Symptoms): Normal daily activity is not affected. EHRA III (Severe Symptoms): Normal daily activity is affected. EHRA IV (Disabling Symptoms): Normal daily activity is discontinued.
Work Productivity and Activity Impairment (WPAI) questionnaire | 1 year
  Change in patient-reported outcome as assessed by the Work Productivity and Activity Impairment (WPAI) questionnaire. The WPAI questionnaire is interpreted by calculating four key impairment percentages over the past 7 days, with higher scores (0-100%) indicating greater impairment and lower productivity. It measures absenteeism (time missed), presenteeism (impairment while working), overall work loss, and daily activity impairment, using a 0-10 scale for productivity.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 12 months after publication
Access Criteria: Upon reasonable request to the Principal Investigator